CLINICAL TRIAL: NCT03997630
Title: Post Traumatic Early Use of High Flow Oxygenation Versus Standard Oxygen for Management of Moderately Hypoxemic Thoracic Trauma: TrOMaTho Study
Brief Title: Management of Moderately Hypoxemic Thoracic Trauma
Acronym: TrOMaTho
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC18.0159
Record Dates: First submitted 2019-03-26; First posted 2019-06-25 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chest Trauma; High Flow Oxygenation
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Interventional group: All patients included in this group will receive a continuous heated and humidified high-flow (30 to 60 l/min) oxygenation with a nasal cannula for 48 hours. Initially, flow rate will be started at 50 l/min with a FiO2 at 50%. According to the protocol, flow rate and FiO2 will be titrated on SpO2 and respiratory tolerance. Weaning and failure of high-flow oxygenation are described in detail in the study protocol.
  Interventions: Device: High flow Oxygenation
- Control group (Active Comparator): Control group: All patients included in this group will receive a low flow oxygenation (flow rate < 15 l/min) with nasal cannula (flow rate ≤ 6 l/min) or non-rebreathing mask (flow rate ≥ 7 l/min).
  Interventions: Device: Standard oxygen

INTERVENTIONS:
Device: High flow Oxygenation — Interventional group: All patients included in this group will receive a continuous heated and humidified high-flow (30 to 60 l/min) oxygenation with a nasal cannula for 48 hours. Initially, flow rate will be started at 50 l/min with a FiO2 at 50%. According to the protocol, flow rate and FiO2 will be titrated on SpO2 and respiratory tolerance. Weaning and failure of high-flow oxygenation are described in detail in the study protocol.
  Arms: Interventional group
Device: Standard oxygen — Control group: All patients included in this group will receive a low flow oxygenation (flow rate < 15 l/min) with nasal cannula (flow rate ≤ 6 l/min) or non-rebreathing mask (flow rate ≥ 7 l/min).
  Arms: Control group

SUMMARY:
In France, the average incidence of thoracic trauma is 10,000 to 15,000 each year. These patients are at risk of early and late post traumatic respiratory complications as follows: pneumonia, Acute Respiratory Distress Syndrome (ARDS), hypoxemia. Main issues of thoracic trauma management were recently published by French anesthesiologist and intensivist experts. Non-invasive ventilation (NIV) was recommended in case of severe hypoxemia (PaO2/FiO2 < 200). In comparison to conventional oxygenation or mechanical ventilation, NIV reduced length of stay, incidence of complications and mortality in case of severe hypoxemia. For mild or moderate hypoxemic patients, no devices were tested to prevent respiratory complications. At the moment, low-flow oxygenation is administered to these patients in the absence of severe hypoxemia. Recently, many studies have found promising results with high-flow oxygenation delivered by nasal cannula. This device has many physiological advantages: wash out the naso-pharyngeal dead space, increase end expiratory lung volume, deliver a moderate or low level of Positive end-expiratory pressure (PEEP), improve work of breathing and confort. Several randomized controlled trials tested this device in many clinical settings, but there are no studies on its use after thoracic trauma. A comparative trial is needed to evaluate early prophylactic administration of high-flow oxygenation after thoracic trauma.

DETAILED DESCRIPTION:
TrOMaTho study is an investigator-initiated, randomized, unblinded, controlled trial. The aim of this study is to compare a prophylactic use of high-flow nasal cannula oxygenation (experimental group) to low-flow oxygenation (control group) after thoracic trauma. 770 patients will be included. Randomization will be conducted with random block and patients will be randomized in 1:1 ratio in one of the two groups. Randomization process will be stratified on: age (more or less 65 years old), use of peridural analgesia and existence of extra thoracic trauma. Only the oxygenation technique is studied, all other aspects of management will be handle by the attending physician.

All patients will be followed from enrollment to hospital discharge. To ensure the same data collection in all centers, six visits are planned: day (D) 1 (inclusion), D7, D14, D28.

Classical blinded methods cannot be used for the evaluation of these kinds of devices. To ensure the same evaluation for all patients and in all centers, all relevant outcomes will be evaluated by an independent clinical event committee. Statistical analysis will be performed by an independent statistician.

Primary endpoint will be analyzed according to intention to treat. Secondary outcomes will be analyzed as exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (age ≥ 18 years),
* Admitted to intensive care unit for less than 48 hours for the management of chest trauma.
* Closed chest trauma, non-penetrating, with a TTSS score> or equal to 4.
* Need for conventional oxygen therapy to maintain SpO2 greater than or equal to 95%.
* Patient affiliated or beneficiary of a social security scheme
* Patient having signed a consent

Exclusion Criteria:

* Severe hypoxemia defined as a PaO2/FiO2 ratio < 200 noted before randomization
* Recommended indication for NIV: cardiogenic pulmonary oedema, decompensated COPD.
* Indication to immediate oro-tracheal intubation. (will not be excluded patients requiring general anaesthesia for a surgical procedure for a peripheral surgical procedure or embolization)

  * Patient with acute respiratory distress, whatever the cause.
  * Hemodynamic instability marked by a fall of the PAS> 30% or a PAS <110 mmHg despite the initial resuscitation measures
  * Neurological degradation with Glasgow score less than 12
* Pregnant or lactating woman
* Patient under guardianship or curatorship
* Contraindication to the use of one or both devices studied (decaying facial trauma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
safety event | Day 28
  The primary endpoint is a composite endpoint defined by:
  * The use of non-invasive ventilation whatever the cause before the 14th day following the trauma (yes/no) OR
  * The use of orotracheal intubation whatever the cause before the 14th day following on the thoracic traumatism.(yes/no) OR
  * The death any cause confused with D28. (yes/no)

SECONDARY OUTCOMES:
Severe hypoxemia | day 7
  Severe hypoxemia before day 7: SpO2 < 92% or PaO2/FiO2 < 200 without oxygenation
Severe hypoxemia | day 14
  Severe hypoxemia before day 14: SpO2 < 92% or PaO2/FiO2 < 200 without oxygenation
Respiratory tract infection | day 7
  Respiratory tract infection before day 7 defined according to international recommendations on health-associated pneumonia or trachea-bronchitis.
Respiratory tract infection | day 14
  Respiratory tract infection before day 14 defined according to international recommendations on health-associated pneumonia or trachea-bronchitis.
Mechanical ventilation | day 7
  Need for mechanical ventilation before day 7. Criteria used to define the need of mechanical ventilation is an acute respiratory distress defined as: the inability to clear tracheal secretion, a deterioration of neurological status (decrease in GCS of 2 points), a respiratory acidosis (pH < 7,25 and PaCO2 > 45 mmHg), signs of persisting or worsening respiratory failure (respiratory rate > 35/min, high respiratory-muscle workload) with a poor response to another oxygenation device.
Mechanical ventilation | day 14
  Need for mechanical ventilation before day 14. Criteria used to define the need of mechanical ventilation is an acute respiratory distress defined as: the inability to clear tracheal secretion, a deterioration of neurological status (decrease in GCS of 2 points), a respiratory acidosis (pH < 7,25 and PaCO2 > 45 mmHg), signs of persisting or worsening respiratory failure (respiratory rate > 35/min, high respiratory-muscle workload) with a poor response to another oxygenation device.
oxygen free days | day 14
  number of day without oxygen
ventilator free days | day 14
  number of day without ventilation
ICU length of stay | day 90
  number of day in ICU
Hospital length of stay | day 90
  number of day of the total stay in hospital
All cause of mortality | day 28 or day 90
  Mortality (yes/no)
quality of life 3 months after High flow oxgenation with the The Short Form (36) Health Survey score | day 90
  SF 36 questionnary total score
Severity of dyspnea using a Saint Georges respiratory questionnaire | day 90
  Saint Georges questionnary total score

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - Centre Hospitalier de Cornouaille, Quimper, Brittany Region
  - Angers university hospital, Angers
  - CHU de Brest, Brest
  - Chartres Hospital, Chartres
  - HIA Percy, Clamart
  - Dreux hospital, Dreux
  - Le Mans hospital, Le Mans
  - Centre Hospitalier de Bretagne Sud, Lorient
  - La Timone Hospital (AP-HM), Marseille
  - Marseille university horpital, Marseille
  - CHRU de Montpellier, Montpellier
  - Morlaix hospital, Morlaix
  - Nantes university hospital, Nantes
  - CHRU de la Pitié-Salpétrière, Paris
  - Kremlin Bicêtre university hospital (APHP), Paris
  - Rennes, university Hospital, Rennes
  - Tours university hospital, Tours
  - CHBA de Vannes, Vannes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.